CLINICAL TRIAL: NCT03791255
Title: Clinical and Radiographic Evaluation of Light Cured Resin Modified Calcium Silicate Versus Light Cured Calcium Hydroxide in Indirect Pulp Treatment of Primary Molars
Brief Title: Light Cured Resin Modified Calcium Silicate Versus Light Cured Calcium Hydroxide in Indirect Pulp Treatment of Primary Molars
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Ashraf Elbanna, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Indirect pulp primary molars
Record Dates: First submitted 2018-12-27; First posted 2019-01-02 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Deep Carious Lesion; Indirect Pulp Treatment
Keywords: resin modified calcium silicate; indirect pulp treatment; primary molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin Modified Calcium Silicate (Experimental): light-cured resin-modified calcium silicate-filled base/ liner material designed for direct and indirect pulp capping
  Interventions: Drug: Calcium silicate liner
- Light Cured Calcium Hydroxide (Active Comparator): gold standard for pulp capping, It allows for the formation of a reparative dentine bridge through cellular differentiation, extracellular matrix secretion and subsequent mineralization.
  Interventions: Drug: Calcium hydroxide liner

INTERVENTIONS:
Drug: Calcium silicate liner — new light-cured resin-modified calcium silicate-filled base/ liner material designed for direct and indirect pulp capping
  Arms: Resin Modified Calcium Silicate
Drug: Calcium hydroxide liner — Calcium hydroxide is the gold standard for pulp capping, allows for the formation of a reparative dentin bridge
  Arms: Light Cured Calcium Hydroxide

SUMMARY:
The objective of this study is to explore if light cured resin modified Calcium silicate could result in better clinical and radiographic success if compared to light cured Calcium hydroxide when used in indirect pulp capping treatment in primary molars.

DETAILED DESCRIPTION:
To evaluate clinical and radiographic success of resin modified calcium silicate in comparison to light cured calcium hydroxide as indirect pulp capping materials in primary molars.

P: Children aged (4-7 years) with deep carious lesions in lower primary second molars indicated for indirect pulp treatment.

I: Indirect pulp treatment using light cured resin modified Calcium Silicate (TheraCal).

C: Indirect pulp treatment using light cured Calcium Hydroxide. O: clinical and radiographic success.

ELIGIBILITY:
Inclusion Criteria:

1. Medically free children.
2. Age range from 4-7 years.
3. Presence of lower second primary molars with deep carious occlusal lesion.
4. No history of spontaneous pain (reversible pulpitis).
5. Clinically: Absence of swelling, sinus, fistula, pain on percussion and tooth mobility.
6. Radiographically: Absence of radiolucent lesions at furcation or periapical region and absence of internal or external root resorption.

Exclusion Criteria:

1. Uncooperative children.
2. Any unmet previous criterion.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 1 month
  Pain questionnaire (binary yes/no)
Postoperative pain | 3 months
  Pain questionnaire (binary yes/no)
Postoperative pain | 6 months
  Pain questionnaire (binary yes/no)
Postoperative pain | 12 months
  Pain questionnaire (binary yes/no)

SECONDARY OUTCOMES:
Swelling | 1 month
  Visual examination by the operator (binary yes/no)
Swelling | 3 months
  Visual examination by the operator (binary yes/no)
Swelling | 6 months
  Visual examination by the operator (binary yes/no)
Swelling | 12 months
  Visual examination by the operator (binary yes/no)
Sinus or fistula | 1 month
  Visual examination by the operator (binary yes/no)
Sinus or fistula | 3 months
  Visual examination by the operator (binary yes/no)
Sinus or fistula | 6 months
  Visual examination by the operator (binary yes/no)
Sinus or fistula | 12 months
  Visual examination by the operator (binary yes/no)
Tooth mobility | 1 month
  back of the mirror to check mobility (binary yes/no)
Tooth mobility | 3 months
  back of the mirror to check mobility (binary yes/no)
Tooth mobility | 6 months
  back of the mirror to check mobility (binary yes/no)
Tooth mobility | 12 months
  back of the mirror to check mobility (binary yes/no)
pain on percussion | 1 month
  back of the mirror to check pain on percussion (binary yes/no)
pain on percussion | 3 months
  back of the mirror to check pain on percussion (binary yes/no)
pain on percussion | 6 months
  back of the mirror to check pain on percussion (binary yes/no)
pain on percussion | 12 months
  back of the mirror to check pain on percussion (binary yes/no)
Occurrence of radiolucent lesions at furcation or periapical region | 1 months
  (binary yes/no)
Occurrence of radiolucent lesions at furcation or periapical region | 3 months
  (binary yes/no)
Occurrence of radiolucent lesions at furcation or periapical region | 6 months
  (binary yes/no)
Occurrence of radiolucent lesions at furcation or periapical region | 12 months
  (binary yes/no)
widening in the periodontal membrane space | 1 month
  (binary yes/no)
widening in the periodontal membrane space | 3 months
  (binary yes/no)
widening in the periodontal membrane space | 6 months
  (binary yes/no)
widening in the periodontal membrane space | 12 months
  (binary yes/no)
presence of internal or external root resorption | 1 month
  (binary yes/no)
presence of internal or external root resorption | 3 months
  (binary yes/no)
presence of internal or external root resorption | 6 months
  (binary yes/no)
presence of internal or external root resorption | 12 months
  (binary yes/no)

IPD SHARING:
Plan to Share IPD: No